CLINICAL TRIAL: NCT00011310
Title: Cardiopulmonary Effects of Particulate Exposure
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9860-CP-001
Record Dates: First submitted 2001-02-15; First posted 2001-02-19 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Respiratory Tract Diseases; Cardiac Diseases; Bronchitis
Keywords: Particulates; Air Pollution; Cardiopulmonary Disease; Lung; Inflammation
MeSH Terms: conditions — Respiratory Tract Diseases; Heart Diseases; Bronchitis; Pulmonary Heart Disease; Inflammation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The aim of this study is to assess cardiac rate and respiratory responses and rhythm after workplace exposure to combustion particulates. A repeated measurement study is being performed on acute boilermakers (apprentices and journeymen). A stratified analysis is then done on those with and without chronic bronchitis, after adjustment for relevant covariates.

DETAILED DESCRIPTION:
Population-based epidemiologic studies of communities in the United States have revealed a consistent association between ambient particulate air pollution and increases in morbidity and mortality. The observed increases result from both respiratory and cardiovascular diseases. Similar associations have been observed for rates of hospital admissions for respiratory and cardiovascular diseases for subjects over age 65. These ambient exposures are to low levels of particulates, many times lower than occupational exposures faced by workers in a variety of industries, including manufacturing, construction, transportation and electric-power generation. The objective of this proposal is to investigate the role of occupational exposure to particulates in the development of respiratory and cardiac responses in boilermakers. We will employ a detailed, continuous-exposure assessment to PM2.5 with repeated measures of biologic and physiologic markers of response. Specific hypotheses to be tested will include: (1) occupational exposure to fuel-oil ash particulates induce airway inflammation as reflected in increased expired NO, and airflow obstruction as reflected in decreases in peak flow (PEFR) and FEV1; (2) particulate exposure will result in acute changes in cardiovascular function, as reflected in changes in heart rate, heart-rate variability and blood pressure; (3) particulate exposures result in increased serum fibrinogen levels, a known risk factor for cardiovascular disease; and (4) chronic bronchitis predisposes particulate-exposed workers to changes in cardiac function. The results of this study will have important implications for preventive efforts aimed at reducing morbidity and mortality from occupational exposure to respirable particulates.

ELIGIBILITY:
Adults; Over 18; Boilermakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Study Completion 2002-02

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard School of Public Health, Boston, Massachusetts, United States